CLINICAL TRIAL: NCT03770702
Title: Investigational and Comparative Study Between the Anti-inflammatory Effectof Both Angiotensin Reeptor Blockers and Statins on Rheumatoid Arthritis Disease Activity on Egyptian Patients
Brief Title: Statins and ARBs on Rheumatoid Activity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rheumatoid
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Angiotensin Receptor Antagonists; Hydroxymethylglutaryl-CoA Reductase Inhibitors; ORANGE protein, Arabidopsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): No intervention
- Angiotensin receptor blockers (Active Comparator): ARB ( Angiotensin receptor blockers) + Traditional therpy.
  Interventions: Drug: Angiotensin receptor blockers
- Statins (Active Comparator): Statin + Traditional therapy.
  Interventions: Drug: Statins

INTERVENTIONS:
Drug: Angiotensin receptor blockers — Candesartan
  Other Names: Cansartan
  Arms: Angiotensin receptor blockers
Drug: Statins — Atorvastatin
  Other Names: Ator
  Arms: Statins

SUMMARY:
Investigational and comparative study between the anti-inflammatory effectof both angiotensin reeptor blockers and statins on rheumatoid arthritis disease activity on Egyptian patients

DETAILED DESCRIPTION:
The study aims at ivestigating and comparing the anti-inflammatory effectof both angiotensin reeptor blockers and statins on rheumatoid arthritis disease activity on Egyptian patients

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis.

Exclusion Criteria:

* Pregnant or lactating
* Hepatic or renal impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in disease activity score | 6 months
  DAS28-ESR

CONTACTS AND LOCATIONS:
Overall Officials: Sahar K Hegazy, Prof, Principal Investigator — Head of Clinical Pharmacy Department; Tarek M Mostafa, Prof, Study Director — Prof of Clinical Pharmacy; Emad M Elshebini, MD, Study Chair — Rheumatology Dept. - Menoufia University; Ahmed HM El-Abd, Msc, Study Chair — Clinical pharmacy Department-Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided